CLINICAL TRIAL: NCT05804305
Title: Misoprostol for Non-alcoholic Steatohepatitis- a Randomized Control Trial
Brief Title: Misoprostol for NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Collaborators: Nabiqasim Industries (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, DR MEHREEN SIYAL, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3280221MSGE
Record Dates: First submitted 2023-01-20; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: NASH
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: This is a double blind randomised control trial to see the effect of Misoprostol in treating patients with NASH
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol (Active Comparator): 600 mcg of Misoprostol per day in three divided doses was given to the patients in the treatment group for a period of two months
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Placebo was given to the patients three times daily for a duration of two months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Misoprostol is a prostaglandin E1 analogue
  Arms: Misoprostol
Drug: Placebo — Placebo contained substance that has no therapeutic value.
  Arms: Placebo

SUMMARY:
The aim of this randomised control trial is to evaluate the effect of Misoprostol in treating patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between age 25 and 64 years
2. Patients having NAFLD as evident by a radiologic test like ultrasound/fibroscan/CT scan etc.
3. ALT level of 1.5 times ULN
4. If already known case of NAFLD, then patient should be on stable doses of Vitamin E, oral hypoglycemics or anti-lipidemic drugs, with no change in medication during 6 months prior to recruitment.

Exclusion Criteria:

1. Patients with age less than 18 yrs or more than 80 yrs,
2. Women of childbearing age
3. Clinically significant acute or chronic liver disease unrelated to NAFLD
4. Evidence of hepatitis B and C
5. Evidence of primary biliary cirrhosis, primary sclerosing cholangitis, or biliary obstruction
6. Autoimmune hepatitis
7. Drug-induced steatohepatitis (ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months)
8. Any cardiovascular event or evidence of active CVS disease
9. Type 1 Diabetes
10. Those consuming alcohol of over 20 grams/day for males and 10 grams/day for females
11. Severe end-organ damage
12. Human immunodeficiency virus (HIV) infection
13. Compensated and decompensated cirrhosis
14. Patients with uncontrolled diabetes
15. Mental instability or incompetence

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in liver function tests | Baseline to 2 Months
  The change in serum alanine aminotransferase (ALT) measured in international units per liter (IU/L), aspartate aminotransferase (AST) in IU/L, gamma-glutamyl transferase (GGT) in IU/L, alkaline phosphatase (ALP) in IU/L, total bilirubin in milligrams per decilitre (mg/dl), direct bilirubin in mg/dl and indirect bilirubin in mg/dl from baseline was ascertained by performing paired sample t-test.
Change From Baseline in Interleukin-6 (IL-6) | Baseline to 2 Months
  The change in Interleukin-6 measured in picograms per milliliter (pg/ml) from baseline was ascertained by performing paired sample t-test.
Change From Baseline in endotoxin levels | Baseline to 2 Months
  The change in endotoxin levels measured in endotoxin units per milliliter (EU/mL) from baseline was ascertained by performing paired sample t-test.

SECONDARY OUTCOMES:
Change From Baseline in hepatic steatosis | Baseline to 2 Months
  The change in hepatic fibrosis from baseline, measured in kilopascals (kPa) by doing fibroscan, was ascertained by performing paired sample t-test.
Change From Baseline in hepatic fibrosis | Baseline to 2 Months
  The change in hepatic fibrosis from baseline, measured through the controlled attenuation parameter (CAP) by doing fibroscan, was ascertained by performing paired sample t-test.
Change From Baseline in dyslipidemia | Baseline to 2 Months
  The change in serum cholesterol level measured in mg/dl, triglycerides in mg/dl, HDL (high-density lipoprotein) cholesterol in mg/dl, LDL (low-density lipoprotein) cholesterol in mg/dl, VLDL (very low-density lipoprotein) cholesterol in mg/dl, non-HDL cholesterol in mg/dl, from baseline by doing fasting lipid profile and performing paired sample t-test.
Change From Baseline in Insulin resistance | Baseline to 2 Months
  The change in Insulin resistance as ascertained by measuring fasting insulin in millionths of an International Unit per milliliter(uU/mL), and fasting blood sugar in mg/dl and then calculating homeostasis model assessment-estimated insulin resistance (HOMA-IR).
  HOMA IR calculation formula:
  HOMA IR = fasting insulin (uU/mL) x fasting glucose (mg/dl)/405
Incidence of Adverse Events | Baseline to 2 Months
  Safety and tolerability were measured by providing adverse event form to the study participants. Any adverse event experienced by the study participants was mentioned in the adverse event form and notified to the primary investigator through a phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Mehreen Siyal, MBBS, FCPS-1, Principal Investigator — Dr. Ziauddin Hospital Clifton
Locations (1):
- Dr. Ziauddin Hospital Clifton, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Siyal M, Abbas Z, Qadeer MA, Saeed A, Ali U, Khatoon A. Misoprostol for non-alcoholic steatohepatitis: a randomised control trial. BMJ Open Gastroenterol. 2024 Jun 6;11(1):e001342. doi: 10.1136/bmjgast-2023-001342. PMID 38844374